CLINICAL TRIAL: NCT01217294
Title: Intrathecal Opioid Versus Ultrasound Guided Fascia Iliaca Plane Block for Analgesia After Primary Hip Arthroplasty
Brief Title: Study Comparing a Nerve Block With Spinal Opiate to Provide Pain Relief for Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Kearns (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Rachel Kearns, co-investigator, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN10AN280
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Analgesia
Keywords: anaesthetic techniques, regional; analgesia, post-operative; fascia iliaca compartment block; ultrasound guided; surgery, orthopaedic
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal morphine, sham block (Sham Comparator): Spinal anaesthesia with hyperbaric bupivacaine 10 - 15mg as specified by the anaesthetist performing the spinal injection, and with the addition of intrathecal morphine 100 micrograms. Sham ultrasound guided fascia iliaca plane block with saline.
  Post-operative analgesia with Paracetamol 1g four times daily, and patient controlled analgesia (PCA) with morphine (1mg bolus, 5 minute lockout period)
  Interventions: Procedure: spinal morphine
- ultrasound guided fascia iliaca block (Active Comparator): Spinal anaesthesia with hyperbaric bupivacaine at a dose between 10 and 15mg as deemed appropriate by the anaesthetic doctor performing the spinal injection, no spinal morphine and fascia iliaca plane block using 2mg/kg levobupivacaine diluted to a total of 40ml with sterile saline.
  Post-operative analgesia with Paracetamol 1g four times daily, and patient controlled analgesia (PCA) with morphine (1mg bolus, 5 minute lockout period)
  Interventions: Procedure: ultrasound guided fascia iliaca block

INTERVENTIONS:
Procedure: ultrasound guided fascia iliaca block — Spinal anaesthesia with hyperbaric bupivacaine at a dose between 10 and 15mg as deemed appropriate by the anaesthetic doctor performing the spinal injection, no spinal morphine and ultrasound guided fascia iliaca plane block using 2mg/kg levobupivacaine diluted to a total of 40ml with sterile saline.
  Arms: ultrasound guided fascia iliaca block
Procedure: spinal morphine — Spinal anaesthesia with hyperbaric bupivacaine 10 - 15mg as deemed appropriate by the anaesthetists performing the spinal injection, and with the addition of intrathecal morphine 100 micrograms. Sham fascia iliaca plane injection with saline.
  Arms: spinal morphine, sham block

SUMMARY:
Pain control after hip replacement surgery is important to ensure patient comfort, allow mobilisation, and aid recovery. The investigators propose a simple and pragmatic study comparing two different anaesthetic techniques in the provision of pain relief after hip surgery. Patients will be randomised to receive either spinal anaesthesia containing morphine or spinal anaesthesia without morphine and an ultrasound guided fascia iliaca nerve block. Although morphine is an effective pain killer, its side effects include itch, urinary retention, nausea and potentially fatal breathing problems. If the nerve block can be shown to provide comparable pain relief to spinal morphine, then morphine could be removed from the spinal injection. This could reduce side effects and improve patient safety. The investigators wish to investigate whether ultrasound guided fascia iliaca plane block provides analgesia which is comparable to that of intrathecal opioid for primary hip arthroplasty in the first 24 hours after hip replacement surgery

DETAILED DESCRIPTION:
There were 6312 primary hip replacements performed in Scotland during the one year period 2007 - 2008. Patients undergoing hip arthroplasty commonly have significant comorbidity and associated polypharmacy providing many potential challenges for the anaesthetic doctor. The optimal way to anaesthetise these patients remains to be fully established although many potential methods exist. The main choice is between general anaesthesia (GA) and regional anaesthesia (RA) or a combination of the two. In a recent systematic review, RA was found to reduce post-operative pain, morphine consumption and nausea and vomiting compared with systemic analgesia.

Spinal anaesthesia is a popular form of RA used in many patients undergoing hip arthroplasty. Opioid drugs are frequently added to the spinal injection in order to prolong post-operative pain relief. However, this is associated with side effects including respiratory depression, urinary retention, nausea and vomiting, and pruritus. Such adverse effects may be uncomfortable for the patient and can delay mobilisation, recovery and eventual discharge.

In patients undergoing hip arthroplasty, peripheral nerve blockade has been shown to improve pain scores and reduce morphine consumption. A peripheral nerve block called the fascia iliaca plane block has shown significant promise as a method of providing sensory blockade of the main nerves which supply pain to the hip. The use of ultrasound for the performance of fascia iliaca plane block has been shown to increase reliability compared with the landmark technique though the clinical benefits of this have not yet been fully investigated.

Compared to nerve stimulation or landmark techniques of nerve localisation, ultrasound has been shown to increase success rates, reduce block onset time, increase block duration, reduce volumes of local anaesthetic required and increase patient satisfaction.

The investigators hypothesise that by increasing the success rate of the fascia iliaca block with ultrasound, it will be possible to achieve superior analgesia post-operatively. Our aim is to assess whether the ultrasound guided fascia iliaca plane block can be used as an alternative to intrathecal morphine in the provision of post-operative analgesia for primary hip arthroplasty. If this is the case, intrathecal opioid could be removed from the spinal anaesthetic. This could in theory have significant safety benefits whilst also reducing side effects. Ultrasound guided fascia iliaca block has not yet been evaluated clinically as a method of providing post-operative analgesia following primary hip arthroplasty. The investigators believe that further investigation of this technique will provide a valuable contribution to existing knowledge and will change current practice.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Competent to give consent
* ASA physical status I - III
* 18-85 years of age, inclusive
* 50-110 kg, inclusive
* Scheduled for unilateral primary hip arthroplasty

Exclusion Criteria:

* Contraindications to fascia iliaca plane block
* Contraindication to spinal anaesthesia
* Coagulopathy, malignancy or infection in the inguinal area
* Patient preference for general anaesthesia
* Allergy to opioids
* Significant peripheral neuropathy or neurologic disorder affecting the lower extremity
* Pregnancy
* History of alcohol or drug dependency / abuse
* History of long term opioid intake
* History of significant psychiatric conditions that may affect patient assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be post-operative morphine consumption in a 24 hour period as self-administered using a patient controlled analgesia (PCA) pump. | 24 hours
  We hypothesise that ultrasound guided fasca iliaca plane block provides analgesia which is comparable to that of intrathecal opioid for primary hip arthroplasty in the first 24 hours after surgery. This study is powered to detect a difference of 10mg of morphine within a 24 hour period. We would consider a dose of 10mg as being significant clinically.

SECONDARY OUTCOMES:
Pain scores | 48 hours
  Pain scores at 48 hours as recorded post-operatively on the PCA chart where time zero is the end of the operation (numerical pain rating score 0 - 10 where 0 is no pain and 10 is worst pain imaginable).
Hypotension | 48 hours
  Incidence of hypotension as defined by systolic blood pressure < 80mmHg or a drop of >25% from baseline systolic pressure, or requiring vasopressor in the first 48 hours post-operatively.
post-operative nausea and vomiting | 48 hours
  Incidence of post-operative nausea and vomiting as defined by nausea score of greater than or equal to 2 (on a PONV scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe nausea and 4 = patient vomiting) or requiring the administration of an anti-emetic agent in the first 48 hours post-operatively.
Pruritus | 48 hours
  Incidence of pruritus as defined by itch felt to be distressing by the patient on questioning after the first 48 hour period post-operatively or requiring treatment with naloxone.
Sedation | 48 hours
  Incidence of sedation as defined by sedation score of greater than or equal to 2 (where 0 = awake, S = normal sleep, 1 = drowsy but easy to rouse, 2 = sedated and difficult to rouse, and 3 = unconscious) or requiring naloxone administration in the first 48 hours post-operatively.
Urinary retention | 48 hours
  Incidence of urinary retention as defined by the requirement for urinary catheterisation due to failure to pass urine in the first 48 hours post-operatively.
First mobilisation | 48 hours
  Time to first mobilisation as defined by patient able to mobilise from bed to chair in hours from time zero as recorded by physiotherapy staff.
Patient satisfaction | 48 hours
  Patient satisfaction as measured using a visual analogue scale (VAS) from 0 - 100mm where 0 is absolutely not satisfied and 100 is completely satisfied. This will be performed after 48 hours and at a routine follow up appointment 3 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: John Kinsella, MBBS MD, Principal Investigator — University Section of Anaesthesia, Glasgow University
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Kearns RJ, Macfarlane AJ, Anderson KJ, Kinsella J. Intrathecal opioid versus ultrasound guided fascia iliaca plane block for analgesia after primary hip arthroplasty: study protocol for a randomised, blinded, noninferiority controlled trial. Trials. 2011 Feb 21;12:51. doi: 10.1186/1745-6215-12-51. PMID 21338492